CLINICAL TRIAL: NCT04614753
Title: A Clinical Trial to Determine the Activity of Dealcoholized Muscadine Wine to Alleviate Oxidative Stress, Inflammation, Skin Photoaging, and Alter the Gut Microbiome in Women 40-67
Brief Title: Dealcoholized Muscadine Wine and Skin Health in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB202000789
Record Dates: First submitted 2020-10-20; First posted 2020-11-04 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2024-10

CONDITIONS: Skin Health

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dealcoholized Muscadine Wine (Active Comparator): Participants in this arm will receive 300ml of dealcoholized muscadine wine daily for six weeks. After a 7- day run-in period, participants will receive dealcoholized muscadine wine daily for six weeks
  Interventions: Other: Dealcoholized Muscadine Wine; Other: Control Beverage
- Control Beverage (Active Comparator): Participants in this arm will receive 300 ml of sugar water and acid content for six weeks. After a 7-day run in period, participants will receive sugar water for six weeks.
  Interventions: Other: Dealcoholized Muscadine Wine; Other: Control Beverage

INTERVENTIONS:
Other: Dealcoholized Muscadine Wine — 300 ml of Dealcoholized Muscadine Wine
Other: Control Beverage — 300ml of Sugar Water and Acid Content

SUMMARY:
The objective of this clinical trial is to determine the activity of dealcoholized muscadine wine to alleviate oxidative stress, inflammation, skin photoaging, and alter gut microbiome in women 40-67 years of age. The investigators hypothesize that dealcoholized muscadine wine daily for 42 days will significantly alleviate oxidative stress, inflammation, skin photoaging, and alter the gut microbiome in women compared to drinking sugar water.

DETAILED DESCRIPTION:
Aging of the skin is characterized by wrinkling, sagging, and laxity. About 80% of facial skin aging is classified as extrinsic, or photoaging because it results from exposure to UV light of the sun that causes oxidative stress The remaining 20% of facial aging is the intrinsic type which is partially caused by the accumulation of proteins that are modified by reactive carbonyls in a reaction known as protein glycation. Aging also shifts the composition of the gut microbiome in at least 35 genera towards an unhealthy state of dysbiosis.

Previous studies showed that muscadine polyphenols inhibited protein glycation under a simulated physiological condition. Additional experiments using cell culture and mice showed that dealcoholized muscadine wine alleviated inflammation and protected against dysbiosis in the gut. The objective of this research is to confirm the health benefits of muscadine wine polyphenols in a clinical trial. The investigators hypothesize that dealcoholized muscadine wine consumption in women 40-65 years old will alleviate skin photoaging and skin conditions by decreasing oxidative stress and inflammation. It is also expected to improve the composition of the gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Healthy,
* BMI 20.0-29.9
* Fitzpatrick skin type 2 and 3.

Exclusion Criteria:

* pregnancy
* breast-feeding
* smoking
* alcohol use
* history of skin cancer
* intake of medication that might influence the outcome of the study
* sunbathing or the use of tanning bed
* intake of vitamin/mineral supplements

Ages: 40 Years to 67 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Sensitivity of skin to UV radiation | Baseline, 28 days
  Irradiation will be applied to dorsal skin (back, scapular region not typically exposed to the sun) with 2 times of minimal erythema dose using an FDA approved UVB phototherapy light and a UV light meter. At each time point on day 0 and 29, skin color will be measured before and 24 h after irradiation. Skin color will be evaluated by a colorimeter.

SECONDARY OUTCOMES:
skin transepidermal water loss | Baseline, 28 days
  Skin transepidermal water loss will be measured using a Tewameter (CK Electronic GmbH, Germany) to evaluate the water barrier function of the skin. The Tewameter measures the density gradient of the water evaporation from the skin (g/h/m^2)
Change in Gut Microbiome | Baseline, 28 days
  Fecal samples will be collected and microbial DNA will be extracted from fecal samples . The 16S ribosomal gene (V1-3 region) of each sample will be amplified and sequenced using a barcoding system on a MiSeq sequencer.
skin hydration | Baseline, 28 days
  Skin hydration will be measured with a Corneometer (CK Electronic GmbH, Germany).
skin erythema and melanin index | Baseline, 28 days
  Skin erythema and melanin index will be assessed with Mexameter (CK Electronic GmbH, Germany). These two components are mainly responsible for the color of the skin. They are measured by reflectance.
skin pH | Baseline, 28 days
  Skin pH will be measured using a Skin-pH-Meter (CK Electronic GmbH, Germany).
Skin smoothness, scaliness, and roughness | Baseline, 28 days
  Skin will be scanned using a probe.
Skin net elasticity, viscoelasticity, and biological elasticity | Baseline, 28 days
  Skin will be measured using a probe.

CONTACTS AND LOCATIONS:
Overall Officials: Liwei Gu, PhD, Principal Investigator — University of Florida
Locations (1):
- Food Science and Human Nutrition Department at University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Chen Y, Mu Q, Hu K, Chen M, Yang J, Chen J, Xie B, Sun Z. Characterization of MK(8)(H(2)) from Rhodococcus sp. B7740 and Its Potential Antiglycation Capacity Measurements. Mar Drugs. 2018 Oct 18;16(10):391. doi: 10.3390/md16100391. PMID 30340371
- [Background] Li R, Kim MH, Sandhu AK, Gao C, Gu L. Muscadine Grape (Vitis rotundifolia) or Wine Phytochemicals Reduce Intestinal Inflammation in Mice with Dextran Sulfate Sodium-Induced Colitis. J Agric Food Chem. 2017 Feb 1;65(4):769-776. doi: 10.1021/acs.jafc.6b03806. Epub 2017 Jan 23. PMID 28112913
- [Background] Micallef M, Lexis L, Lewandowski P. Red wine consumption increases antioxidant status and decreases oxidative stress in the circulation of both young and old humans. Nutr J. 2007 Sep 24;6:27. doi: 10.1186/1475-2891-6-27. PMID 17888186
- [Background] Heinrich U, Moore CE, De Spirt S, Tronnier H, Stahl W. Green tea polyphenols provide photoprotection, increase microcirculation, and modulate skin properties of women. J Nutr. 2011 Jun;141(6):1202-8. doi: 10.3945/jn.110.136465. Epub 2011 Apr 27. PMID 21525260
- [Background] Heinrich U, Neukam K, Tronnier H, Sies H, Stahl W. Long-term ingestion of high flavanol cocoa provides photoprotection against UV-induced erythema and improves skin condition in women. J Nutr. 2006 Jun;136(6):1565-9. doi: 10.1093/jn/136.6.1565. PMID 16702322
- [Background] Heckman CJ, Chandler R, Kloss JD, Benson A, Rooney D, Munshi T, Darlow SD, Perlis C, Manne SL, Oslin DW. Minimal Erythema Dose (MED) testing. J Vis Exp. 2013 May 28;(75):e50175. doi: 10.3791/50175. PMID 23748556